CLINICAL TRIAL: NCT06039501
Title: The Family Perspectives Project Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Modes (Other)
Collaborators: National Palliative Care Research Center (Other)
Responsible Party: Sponsor-Investigator, Matthew Modes, Assistant Professor, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Study00002813
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Failure; Family Support; Physician-Patient Relations; Critical Illness
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Perspective Program (Experimental): Families of critically ill patients will receive a program designed to enhance equitable communication and emotional support.
  Questionnaires will be completed by primary surrogate decision makers, ICU support counselors, and ICU care team members (physicians, nurses, social workers). Meetings between families and ICU support counselors will be audio recorded (optional). Meetings between families and ICU care teams will be audio recorded (optional). Interviews with participants will be completed (optional).
  Interventions: Behavioral: Family Perspective Program
- Usual Care (No Intervention): Families of critically ill patients will receive usual care, which involves regular and routine meetings between families and the ICU care team.
  Questionnaires will be completed by primary surrogate decision makers and ICU care team members (physicians, nurses, social workers). Meetings between families and ICU care teams will be audio recorded (optional). Interviews with participants will be completed (optional).

INTERVENTIONS:
Behavioral: Family Perspective Program — The program involves regular meetings between families and an ICU support counselor. The ICU support counselor is a trained expert in providing culturally competent emotional and/or spiritual support. The ICU support counselor will support families and also learn and summarize family perspectives in a standardized report. ICU care team members will be prompted to perspective take as they review reports prior to regular routine meetings between families and the ICU care team.
  Arms: Family Perspective Program

SUMMARY:
The purpose of the study is to conduct a pilot randomized trial of a program designed to enhance equitable communication and emotional support for families of critically ill patients in order to determine feasibility, acceptability, and participant experience with the program.

The primary study procedures include: chart abstraction, questionnaires, meetings with ICU support counselors, meetings with ICU physicians and care team, audio recordings of these meetings (optional), and interviews with study participants (optional).

Study participants include: 70 critically ill patients with acute respiratory failure (enrolled with the consent of their Legally Authorized Representative) and their primary surrogate decision makers as well as ICU support counselors and ICU care teams (physicians, nurses, social workers).

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria:

  * Individuals 18 years old or older.
  * Individuals admitted to the medical intensive care unit (MICU) at Cedars-Sinai Medical Center.
  * Individuals with acute respiratory failure, defined as >24 hours of invasive mechanical ventilation.
  * Individuals who received invasive mechanical ventilation within 24 hours of admission to the MICU.
  * Individuals expected to need invasive mechanical ventilation for >72 hours total, as determined by the patient's intensivist physician (fellow or attending).
* Primary surrogate decision maker inclusion criteria:

  o Individuals 18 years old or older.
  * Individual who self-identifies as the most responsible for making decisions for the enrolled patient (can be either family member or close friend).
  * Proficiency in English language.
* ICU support counselor inclusion criteria:

  * Individuals 18 years old or older.
  * Individuals who work as hospital chaplains in the MICU.
* Physician (intensivist) inclusion criteria:

  * Individuals 18 years old or older.
  * Individuals who work as critical care physicians in the MICU (fellow or attending).
* Nurse inclusion criteria:

  * Individuals 18 years old or older.
  * Individuals who work as bedside nurses in the MICU.
* Social worker inclusion criteria:

  * Individuals 18 years old or older.
  * Individuals work as social workers in the MICU.

Exclusion Criteria:

* Patient exclusion criteria:

  o Any records flagged "break the glass" or "research opt out."

  o Individuals expected to die within 24 hours of potential enrollment, as determined by the patient's intensivist physician (fellow or attending).

  o Individuals on comfort care protocol or with clear preference for comfort care, as determined by the patient's intensivist physician (fellow or attending).
  * Individuals who are chronically dependent on a ventilator prior to admission.
  * Individuals with acute on chronic neuromuscular disease-related respiratory failure (e.g., Guillain Barre, Muscular Dystrophy, Myasthenia Gravis, etc.).
  * Individuals imminently awaiting organ transplant, as determined by the patient's intensivist physician (fellow or attending).
  * Individuals with decisional capacity, as determined by the patient's intensivist physician (fellow or attending).
  * Individuals who are unrepresented (i.e., patient has no surrogate decision maker).
  * Individuals whose potential enrolled family member (primary surrogate decision maker) is not proficient in English.
  * Individuals whose attending physician is the PI on this study at the time of potential enrollment.
  * Individuals who are cared for by intensivist physicians (fellow and attending) who do not agree to participate in the study.
  * Individuals who have a pre-existing relationship with a hospital chaplain who does not agree to participate in the study, as determined by that chaplain.
* Primary surrogate decision maker exclusion criteria:

  o Not proficient in English language. (Rationale: materials and intervention are not adapted in other languages.)
* ICU support counselor exclusion criteria:

  o None
* Physician (intensivist) exclusion criteria:

  o None
* Nurse exclusion criteria:

  o None
* Social worker exclusion criteria:

  * None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the program for families of patients with acute respiratory failure. | 6 months
  The proportion of enrolled primary surrogate decision makers randomized to the program who receive all program components. The study will be declared "feasible" if at least 70% of primary surrogate decision makers receive all program components (meeting with ICU support counselors, ICU support counselors generating standardized reports, reports being reviewed by ICU care team members prior to meeting with families).

SECONDARY OUTCOMES:
Feasibility of collecting data from families | 6 months
  The proportion of enrolled primary surrogate decision makers completing all questionnaires (enrollment, after meetings with ICU care team, 1-month post-enrollment, and 6 months post-enrollment) in each arm.
Feasibility of collecting data from ICU support counselors | 6 months
  The proportion of questionnaires (enrollment, after each meeting with a primary surrogate decision maker) completed by ICU support counselors.
Feasibility of collecting data from ICU care team members | 6 months
  The proportion of questionnaires (enrollment, after each meeting with a primary surrogate decision maker) completed by ICU care team members (physicians, nurses, social workers) in each arm.
ICU support counselor perception of feasibility of implementing the program | 6 months
  Mean score on the validated 4-item Feasibility of Intervention Measure
ICU care team member perception of feasibility of implementing the program | 6 months
  Mean score on the validated 4-item Feasibility of Intervention Measure

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Modes, MD, MPP, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No